CLINICAL TRIAL: NCT07201415
Title: An Exploratory Study of the Efficacy and Safety of Minimally Invasive Supraporoidal Drainage for Advanced Neovascular Glaucoma
Brief Title: Minimally Invasive Suprachoroidal Drainage for the Treatment of Neovascular Glaucoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250904
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neovascular Glaucoma
Keywords: Neovascular glaucoma; Retinal Vein Occlusion; Diabetic Retinopathy; Treatment
MeSH Terms: conditions — Glaucoma, Neovascular; Retinal Vein Occlusion; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Treatment Group (Experimental): The patient will undergo a minimally invasive suprachoroidal drainage procedure
  Interventions: Procedure: minimally invasive suprachoroidal drainage

INTERVENTIONS:
Procedure: minimally invasive suprachoroidal drainage — minimally invasive suprachoroidal drainage

SUMMARY:
To explore the efficacy and safety of minimally invasive suprachoroidal drainage for the treatment of advanced neovascular glaucoma

DETAILED DESCRIPTION:
To explore the efficacy and safety of minimally invasive supraporcular drainage in the treatment of advanced neovascular glaucoma, and to record the various basic diseases, ocular conditions, lifestyle, inflammatory markers and other parameters of NVG patients. To compare the safety and efficacy of new surgical methods and traditional surgical methods in order to find an effective treatment for neovascular glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Advanced (angle-closure) neovascular glaucoma with poorly controlled intraocular pressure (IOP > 21mmHg) after medical or surgical treatment

Exclusion Criteria:

* Various other types of glaucoma (including primary open-angle glaucoma, primary open-closed glaucoma, normal tension glaucoma, juvenile glaucoma, congenital glaucoma, other special types of glaucoma, etc.)
* Eye infection within two weeks before surgery
* Non-glaucomatous intraocular diseases that affect intraocular pressure (choroidal hemorrhage or detachment, retinal detachment, lens subluxation, thyroid eye disease, clinically significant macular edema, eye tumors, etc.)
* Visual acuity of non-study eyes < 0.05
* Congenital or acquired factors lead to ciliary body anatomical abnormalities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Ocular biological parameters | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  intraocular pressure
Ocular biological parameters | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  visual acuity
Surgical outcome measures | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  use of intraocular pressure lowering drugs
The success rate of surgery was evaluated according to the specific value of intraocular pressure after surgery | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  Complete success was defined as IOP within the normal range with no drug dependence, conditional success was defined as IOP within the normal range with drug dependence, and failure was defined as the rest

SECONDARY OUTCOMES:
The effective rate of surgery was evaluated according to the amplitude of IOP reduction after surgery and the change in the number of IOP-lowering drugs | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  Amplitude of IOP reduction: IOP change/initial IOP.The total number of IOP lowering drugs was recorded based on the number of active ingredients
Surgical outcome measures | 1 day, 1 week, 1 month, 3 months, and 6 months after surgery
  complications

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China